CLINICAL TRIAL: NCT06033690
Title: Intervention Beyond Multidisciplinarity in the Surgical Treatment of Obesity Randomized Clinical Trial
Brief Title: Intervention in the Surgical Treatment of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UP5815/20
Record Dates: First submitted 2023-06-21; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Obesity, Morbid
Keywords: obesity; bariatric surgery; food guide; interdisciplinarity
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: the two groups were randomized by online program, into intervention group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- multidisciplinary guide (Experimental): Consultation and multidisciplinary guide with guidance on physical activity and healthy eating.
  Interventions: Behavioral: multidisciplinary guide
- Control (No Intervention): Consultations with a multidisciplinary team

INTERVENTIONS:
Behavioral: multidisciplinary guide — use of the food guide for education, clarification of doubts
  Arms: multidisciplinary guide

SUMMARY:
The worldwide prevalence of obesity reaching epidemic levels, and directly associated with several non-communicable chronic diseases, being considered the sixth leading cause of death in the world. In Brazil, estimated that one third of the population is overweight. Currently, bariatric surgery the fastest and most effective method to control the disease. However, most patients do not follow the postoperative follow-up protocol, causing weight regain. Intervention in the literature that goes beyond multidisciplinary and can prevent weight relapse. The develop and apply an interdisciplinary manual, based on the guidelines of the Food Guide for the Brazilian Population, as a support in the prophylactic treatment of weight relapse patients and bariatric surgery

DETAILED DESCRIPTION:
The objective of this randomized clinical study is to compare the eating behavior of obese participants who underwent the dietary guide after bariatric surgery treatment. The main questions are:

* Can an interdisciplinary intervention through a dietary guide promote a change in eating behavior in participants undergoing surgical treatment for obesity?
* Participants will participate in consultations and receive a food guidance guide and lectures with guidance.
* Researchers will compare intervention and control groups to see if there will be changes in eating behavior

ELIGIBILITY:
Inclusion criteria:

Referred for bariatric surgery Having or not comorbidity associated with obesity.

Exclusion criteria:

not signing the informed consent form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
behavior | 40 minutes
  participants' scores in a pre- and post-intervention food assessment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Izabele Vian, Study Director — Cardiology Institute
Locations (1):
- Izabele Vian, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No